CLINICAL TRIAL: NCT00003195
Title: A Phase II Study of Total Marrow Irradiation, Busulfan, and Alpha-Interferon Followed by Allogeneic Peripheral Blood Stem Cell or Marrow Transplantation for Treatment of Patients With Advanced Multiple Myeloma.
Brief Title: Total-Body Irradiation, Busulfan, and Interferon Alfa Followed by Peripheral Stem Cell or Bone Marrow Transplantation in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1272.00; FHCRC-1272.00; NCI-H98-0009; CDR0000066030 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Interferon-alpha; Busulfan; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: busulfan
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage cancer cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Interferon alfa may interfere with the growth of cancer cells.

PURPOSE: Phase II trial to study the effectiveness of total-body irradiation, busulfan, and interferon alfa followed by peripheral stem cell or bone marrow transplantation in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the effects of total marrow irradiation and busulfan followed by allogeneic peripheral blood stem cell or marrow transplantation on the outcomes of treatment related mortality, response, relapse, survival, and event free survival for patients with advanced multiple myeloma.

OUTLINE: Peripheral blood stem cell (PBSC) or bone marrow (BM) collection and infusion are performed according to standard practice. Patients undergo total marrow irradiation (TMI) bid for 3 days. Busulfan is administered every 6 hours on days -6 to -3. PBSC or BM is infused on day 0. Interferon alfa is administered subcutaneously on Mondays, Wednesdays, and Fridays beginning on day 80. Interferon therapy may continue in the absence of graft versus host disease or disease progression. Patients are followed on days 56 and 84, then every 6 months for 2 years, and annually thereafter.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued over 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically diagnosed stage II or III multiple myeloma Stage I multiple myeloma progressing on conventional therapy HLA matched donor Related - ages 18-65 Unrelated - ages 18-55

PATIENT CHARACTERISTICS: Age: 18 to 65 Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: No significant hepatic disease Bilirubin no greater than 2 mg/dL Renal: Creatinine clearance at least 40 mL/min Calcium no greater than 15 mg/dL Cardiovascular: No significant cardiac disease Ejection fraction at least 40% Pulmonary: No significant pulmonary disease FEV1 at least 50% OR DLCO at least 50% Other: No obesity Chest wall no greater than 3 cm thick No pendulous breasts HIV negative

PRIOR CONCURRENT THERAPY: Must have received prior conventional therapy for stage I disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-12; Study Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William I. Bensinger, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States